CLINICAL TRIAL: NCT01506141
Title: An Open-Label Extension of Study HGT-HIT-045 Evaluating Long-Term Safety and Clinical Outcomes of Intrathecal Idursulfase-IT Administered in Conjunction With Intravenous Elaprase® in Pediatric Patients With Hunter Syndrome and Cognitive Impairment
Brief Title: An Extension Study of HGT-HIT-045 Evaluating Long-Term Safety and Clinical Outcomes of Idursulfase-IT in Conjunction With Elaprase in Pediatric Participants With Hunter Syndrome and Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-HIT-046; 2011-000212-25 (EudraCT Number)
Record Dates: First submitted 2011-12-15; First posted 2012-01-09 (Estimated); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hunter Syndrome
Keywords: MPS II; MPS 2; lysosomal storage disorder; mps symptoms; enlarged adenoids; elaprase; hunter's syndrome; MPS2; hunters disease; hunter's disease treatment; hunter syndrome therapy; iduronate sulfatase; mps society; MPSII; hunter syndrome treatment; hunter's disease; iduronate 2 sulfatase; mucopolysaccharides; mps diagnosis; chronic ear infection; hunters syndrome; ert treatment; lysosomal storage disease; hunter disease; enzyme replacement therapy; idursulfase; hunter's syndrome treatment
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death; Lysosomal Storage Diseases | interventions — idursulfase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Idursulfase-IT 1 milligram (mg) (Experimental): Participants will receive 1 mg idursulfase-IT intrathecally via intrathecal drug delivery device (IDDD) or lumbar puncture (LP) once monthly and standard-of-care (SoC) therapy of Elaprase intravenous (IV) infusions.
  Interventions: Drug: Idursulfase-IT; Drug: Elaprase
- Idursulfase-IT 10 mg (Experimental): Participants will receive 10 mg idursulfase-IT intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions.
  Interventions: Drug: Idursulfase-IT; Drug: Elaprase
- Idursulfase-IT 30 mg (Experimental): Participants will receive 30 mg idursulfase-IT intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions.
  Interventions: Drug: Idursulfase-IT; Drug: Elaprase

INTERVENTIONS:
Drug: Idursulfase-IT — Idursulfase-IT once monthly via IDDD.
Drug: Elaprase — Weekly IV infusions of commercially available Elaprase.

SUMMARY:
This extension study of HGT-HIT-045 is designed to collect long-term safety data in pediatric participants with Hunter syndrome and cognitive impairment who are receiving intrathecal (IT) idursulfase-IT and intravenous (IV) Elaprase enzyme replacement therapy.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Participant must have completed all study requirements and End of study (EOS) assessments for study HGT-HIT-045 (NCT00920647) prior to enrolling in Study HGT-HIT-046 and must have no safety or medical issues that contraindicate participation.
* The participant's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the participant's parent(s) or legally authorized guardian(s) and the participant's assent, as relevant, must be obtained.
* The participant has received and tolerated a minimum of 12 months of treatment with weekly IV infusions of Elaprase and has received 80% of the total planned infusions within the last 6 months.

Exclusion Criteria:

* The participant is enrolled in another clinical study that involves clinical investigations or use of any investigational product (drug or device) other than the PORT-A-CATH IDDD within 30 days prior to study enrollment or at any time during the study.
* The participant is unable to comply with the protocol (eg, is unable to return for safety evaluations, or is otherwise unlikely to complete the study) as determined by the investigator.
* The participant has experienced an adverse reaction to study drug in Study HGT-HIT-045 (NCT00920647) that contraindicates further treatment with intrathecal idursulfase-IT.
* The participant has a known hypersensitivity to any of the components of idursulfase-IT.
* The participant has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to airway compromise or other conditions.
* The participant has a condition that is contraindicated as described in the SOPH-A-PORT Mini S IDDD Instructions for Use, including:

  1. The participant has had, or may have, an allergic reaction to the materials of construction of the SOPH-A-PORT Mini S device
  2. The participant's body size is too small to support the size of the SOPH-A-PORT Mini S Access Port, as judged by the investigator
  3. The participant's drug therapy requires substances known to be incompatible with the materials of construction
  4. The participant has a known or suspected local or general infection
  5. The participant is at risk of abnormal bleeding due to a medical condition or therapy
  6. The participant has one or more spinal abnormalities that could complicate safe implantation or fixation
  7. The participant has a functioning CSF shunt device
  8. The participant has shown an intolerance to an implanted device

     An additional exclusion criterion for patients who were previously untreated with intrathecal idursulfase-IT in Study HGT-HIT-045 (NCT00920647):
* The participant has an opening CSF pressure upon lumbar puncture that exceeds 30.0 centimeter (cm) water (H2O).

Ages: 3 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (7):
  - Ann & Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Legacy Emanuel Hospital, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Utah Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada
- Birmingham Children's Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Background] Muenzer J, Gucsavas-Calikoglu M, McCandless SE, Schuetz TJ, Kimura A. A phase I/II clinical trial of enzyme replacement therapy in mucopolysaccharidosis II (Hunter syndrome). Mol Genet Metab. 2007 Mar;90(3):329-37. doi: 10.1016/j.ymgme.2006.09.001. Epub 2006 Dec 20. PMID 17185020
- [Background] Muenzer J, Wraith JE, Beck M, Giugliani R, Harmatz P, Eng CM, Vellodi A, Martin R, Ramaswami U, Gucsavas-Calikoglu M, Vijayaraghavan S, Wendt S, Puga AC, Ulbrich B, Shinawi M, Cleary M, Piper D, Conway AM, Kimura A. A phase II/III clinical study of enzyme replacement therapy with idursulfase in mucopolysaccharidosis II (Hunter syndrome). Genet Med. 2006 Aug;8(8):465-73. doi: 10.1097/01.gim.0000232477.37660.fb. PMID 16912578
- [Derived] Muenzer J, Vijayaraghavan S, Stein M, Kearney S, Wu Y, Alexanderian D. Long-term open-label phase I/II extension study of intrathecal idursulfase-IT in the treatment of neuronopathic mucopolysaccharidosis II. Genet Med. 2022 Jul;24(7):1437-1448. doi: 10.1016/j.gim.2022.04.002. Epub 2022 May 20. PMID 35588317
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fce4db2bf003ab46749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites in the United States (US) and the United Kingdom (UK) from 01 August 2010 to 30 April 2024.
Pre-assignment Details: 15 participants who completed the Study HGT-HIT-045 (NCT00920647) received idursulfase-IT in conjunction with Elaprase therapy. Participants who received idursulfase-IT treatment in study HGT-HIT-045, initiated treatment at the same dose level and were analyzed as per the reference timepoints of HGT-HIT-045 for some evaluations. For others, the reference timepoints after enrollment to this extension study were considered.
Groups:
- Idursulfase-IT 10 mg: Participants received 10 mg idursulfase-IT initially intrathecally via intrathecal drug delivery device (IDDD) or lumbar puncture (LP) once monthly and SoC therapy of Elaprase IV infusions up to a maximum of 157.2 months. This included participants who received 1 mg idursulfase-IT initially and then switched to receive 10 mg idursulfase-IT in this arm group after Month 7 or later. These participants were analyzed in this arm group since transition to this group.
- Idursulfase-IT 30 mg: Participants received 30 mg idursulfase-IT intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions for up to a maximum of 148.2 months.
Period: Overall Study
Arm/Group | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Started | 10 | 5
Transferred From 1 mg Arm (Participants received 1 mg idursulfase-IT initially and then switched to 10 mg idursulfase-IT after Month 7 or later.) | 4 | 0
Completed | 3 | 0
Not Completed | 7 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Participation Terminated by Investigator | 1 | 1
Not completed — Site Terminated by Sponsor | 2 | 0
Not completed — Reason Not Specified | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and have had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study. Baseline characteristics are reported according to participant's initial treatment arms.
Groups:
- Idursulfase-IT 1 mg: Participants received 1 mg idursulfase-IT intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions for up to a maximum of 10.1 months.
- Idursulfase-IT 10 mg: Participants received 10 mg idursulfase-IT initially intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions for up to a maximum of 157.2 months.
- Total: Total of all reporting groups
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg | Total
Number analyzed (Participants) | 4 | 6 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.61 (1.799) | 5.68 (2.501) | 7.94 (2.706) | 6.41 (2.502)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 6 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 4 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, and/or laboratory changes occurring in any phase of a clinical trial, and whether or not considered study drug-related. TEAEs were defined as all AEs occurring on or after the first IDDD surgery date or first dose (whichever is earlier) for the participant (whether it is in this extension study or in HGT HIT-045 [NCT00920647]) and before the end of the study (EOS) visit (+30 days). For Idursulfase-IT 1 mg+10 mg arm the summary presented includes only the TEAEs that occurred while the participants were assigned to 10 mg.
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Population: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study.
Measure: Count of Participants; unit: Participants
Groups:
- Idursulfase-IT 10 mg: Participants received 10 mg idursulfase-IT initially intrathecally via IDDD or LP once monthly and SoC therapy of Elaprase IV infusions up to a maximum of 157.2 months. This included participants who received 1 mg idursulfase-IT initially and then switched to receive 10 mg idursulfase-IT in this arm group after Month 7 or later. These participants were analyzed in this arm group since transition to this group.
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
Participants | 4 | 10 | 5

2. Primary Outcome: Number of Participants With Clinically Significant Changes or Apparent Difference Across Treatment Groups in Laboratory Parameters
Description: Number of participants with clinically significant changes in laboratory parameters (chemistry, hematology, urinalysis and CSF values) were collected.
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes or Apparent Difference Across Treatment Groups in 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECG) findings (heart rate, PR interval, QRS interval, QT interval and the corrected QT interval) were collected.
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
Participants | 0 | 0 | 0

4. Primary Outcome: CSF Chemistries: Change From Baseline in CSF Total Cell Count
Time Frame: Baseline, Month 163
Population: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study. Overall number analyzed are the number of participants who had data at Baseline. Number analyzed indicates the number of participants with data available for analyses at specified time points.
Measure: Mean (Standard Deviation); unit: 10^6 cells/Liter (L)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 6 | 5
10^6 cells/Liter (L)
  Baseline | 1.0 (0.00) | 1.0 (0.00) | 1.0 (0.00)
  Change From Baseline in CSF Total Cell Count at Month 163: number analyzed (Participants) | 0 | 3 | 0
  Change From Baseline in CSF Total Cell Count at Month 163 |  | 7.3 (11.85) |

5. Primary Outcome: CSF Chemistries: Change From Baseline in CSF Glucose
Time Frame: Baseline, Month 163
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 6 | 5
millimoles per liter (mmol/L)
  Baseline | 2.950 (0.265) | 2.850 (0.217) | 3.000 (0.200)
  Change from Baseline in CSF Glucose at Month 163: number analyzed (Participants) | 0 | 3 | 0
  Change from Baseline in CSF Glucose at Month 163 |  | 0.523 (0.436) |

6. Primary Outcome: CSF Chemistries: Change From Baseline in CSF Protein
Time Frame: Baseline, Month 163
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 6 | 5
grams per liter (g/L)
  Baseline | 0.400 (0.194) | 0.282 (0.144) | 0.530 (0.368)
  Change from Baseline in CSF Protein at Month 163: number analyzed (Participants) | 0 | 3 | 0
  Change from Baseline in CSF Protein at Month 163 |  | 0.493 (0.229) |

7. Primary Outcome: Number of Participants With Anti-idursulfase Antibodies in CSF
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
Participants
  At Baseline: number analyzed (Participants) | 4 | 6 | 5
  At Baseline | 3 | 1 | 1
  Post-Baseline | 3 | 5 | 1

8. Primary Outcome: Number of Participants With Anti-idursulfase Antibodies in Serum
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
Participants
  At Baseline: number analyzed (Participants) | 4 | 6 | 5
  At Baseline | 3 | 2 | 2
  Post-Baseline | 3 | 6 | 3

9. Secondary Outcome: Area Under the Curve Extrapolated to Infinity (AUC0-infinity) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Area under the curve extrapolated to infinity, calculated using the observed value of the last non-zero concentration (AUC0-infinity) of idursulfase was assessed. Participants in 1 mg arm group were assessed for Pharmacokinetic (PK) analysis in the HGT-HIT-045 study.
Time Frame: 15 minutes prior to IT injection, at 1,2,3,4,6,8,12,24,30,36 hours (±1 hour) following IT injection on Day 2 of Weeks 3,23, for 1 mg arm group and on Day 2 of Weeks 3,23, Months 19,31,43,55,67,79 for 10 and 30 mg arm groups
Population: PK population included all participants who received study drug & participated in the scheduled pharmacokinetic studies,& for whom at least 1 post-dose PK blood sample was collected. Overall number analyzed indicates number of participants with data available for analyses. Number analyzed indicates number of participants with data available for analyses at specified time points.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter(h*ng/mL)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 6 | 5
hours*nanograms per milliliter(h*ng/mL)
  Week 3: Day 2: number analyzed (Participants) | 3 | 0 | 0
  Week 3: Day 2 | NA (NA) — Mean and Standard Deviation (SD) were not estimable as values were below lower limit of quantification (LLOQ). |  |
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 0
  Week 23: Day 2 | 1574.37 (NA) — SD was not estimable for a single participant. | 1765 (NA) — SD was not estimable for a single participant. |
  Month 19: Day 2: number analyzed (Participants) | 0 | 3 | 2
  Month 19: Day 2 |  | 2869 (563.1) | 5179 (2579.8)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 1
  Month 31: Day 2 |  | 2649 (1334.8) | 4766 (NA) — SD was not estimable for a single participant.
  Month 43: number analyzed (Participants) | 0 | 4 | 2
  Month 43 |  | 2324 (203.0) | 4395 (733.1)
  Month 55: number analyzed (Participants) | 0 | 3 | 2
  Month 55 |  | 1636 (351.4) | 2445 (1770.8)
  Month 67: number analyzed (Participants) | 0 | 2 | 2
  Month 67 |  | 1649 (167.4) | 3270 (801.6)
  Month 79: number analyzed (Participants) | 0 | 3 | 0
  Month 79 |  | 1865 (775.2) |

10. Secondary Outcome: Area Under the Curve From the Time of Dosing to the Last Measureable Concentration (AUC0-t) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: PK population included all participants who received study drug and participated in the scheduled pharmacokinetic studies, and for whom at least 1 post-dose PK blood sample was collected. Overall number analyzed indicates the number of participants with data available for analyses. Number analyzed indicates the number of participants with data available for analyses at specified time points.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 7 | 5
h*ng/mL
  Week 3: Day 2: number analyzed (Participants) | 3 | 1 | 1
  Week 3: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. | 1214 (NA) — SD was not estimable for a single participant. | 3746 (NA) — SD was not estimable for a single participant.
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 1
  Week 23: Day 2 | 524.68 (NA) — SD was not estimable for a single participant. | 1047 (NA) — SD was not estimable for a single participant. | 4855 (NA) — SD was not estimable for a single participant.
  Month 19: Day 2: number analyzed (Participants) | 0 | 7 | 5
  Month 19: Day 2 |  | 1633 (976.6) | 3525 (835.5)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 4
  Month 31: Day 2 |  | 2031 (1081.9) | 3586 (1056.9)
  Month 43: number analyzed (Participants) | 0 | 4 | 4
  Month 43 |  | 1944 (295.8) | 3141 (979.7)
  Month 55: number analyzed (Participants) | 0 | 6 | 3
  Month 55 |  | 1356 (235.3) | 1466 (1511.8)
  Month 67: number analyzed (Participants) | 0 | 3 | 3
  Month 67 |  | 1247 (204.0) | 2415 (394.8)
  Month 79: number analyzed (Participants) | 0 | 4 | 0
  Month 79 |  | 1500 (347.1) |

11. Secondary Outcome: Maximum Observed Concentration (Cmax) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 7 | 5
nanograms per milliliter (ng/mL)
  Week 3: Day 2: number analyzed (Participants) | 3 | 1 | 1
  Week 3: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. | 43.95 (NA) — SD was not estimable for a single participant. | 146.75 (NA) — SD was not estimable for a single participant.
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 1
  Week 23: Day 2 | 19 (NA) — SD was not estimable for a single participant. | 36.10 (NA) — SD was not estimable for a single participant. | 173.40 (NA) — SD was not estimable for a single participant.
  Month 19: Day 2: number analyzed (Participants) | 0 | 7 | 5
  Month 19: Day 2 |  | 76.39 (51.386) | 156.80 (33.054)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 4
  Month 31: Day 2 |  | 143.52 (122.774) | 175.20 (70.083)
  Month 43: number analyzed (Participants) | 0 | 4 | 4
  Month 43 |  | 90.57 (28.720) | 144.35 (44.434)
  Month 55: number analyzed (Participants) | 0 | 6 | 3
  Month 55 |  | 61.50 (19.330) | 93.43 (61.406)
  Month 67: number analyzed (Participants) | 0 | 3 | 3
  Month 67 |  | 56.73 (12.690) | 99.20 (19.762)
  Month 79: number analyzed (Participants) | 0 | 4 | 0
  Month 79 |  | 64.08 (7.835) |

12. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of Idursulfase Administered in as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 7 | 5
hours
  Week 3: Day 2: number analyzed (Participants) | 3 | 1 | 1
  Week 3: Day 2 | NA [NA to NA] — Median and Full range were not estimable as values were below LLOQ. | 24.03 [NA to NA] — Full range was not estimable for a single participant. | 36.07 [NA to NA] — Full range was not estimable for a single participant.
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 1
  Week 23: Day 2 | 8.03 [NA to NA] — Full range was not estimable for a single participant. | 12.00 [NA to NA] — Full range was not estimable for a single participant. | 12.00 [NA to NA] — Full range was not estimable for a single participant.
  Month 19: Day 2: number analyzed (Participants) | 0 | 7 | 5
  Month 19: Day 2 |  | 12.00 [6.00 to 36.2] | 24.00 [2.00 to 30.0]
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 4
  Month 31: Day 2 |  | 9.99 [1.12 to 12.0] | 17.98 [6.00 to 30.1]
  Month 43: number analyzed (Participants) | 0 | 4 | 4
  Month 43 |  | 12.00 [8.00 to 12.0] | 10.02 [6.03 to 12.0]
  Month 55: number analyzed (Participants) | 0 | 6 | 3
  Month 55 |  | 12.00 [6.00 to 12.0] | 7.97 [2.00 to 8.00]
  Month 67: number analyzed (Participants) | 0 | 3 | 3
  Month 67 |  | 12.00 [6.00 to 12.0] | 12.00 [6.00 to 30.0]
  Month 79: number analyzed (Participants) | 0 | 4 | 0
  Month 79 |  | 10.00 [8.00 to 12.00] |

13. Secondary Outcome: Total Body Clearance for Extravascular Administration Divided by the Fraction of Dose Absorbed (Cl/F) of Idursulfase-IT Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 6 | 5
liters per hour (L/h)
  Week 3: Day 2: number analyzed (Participants) | 3 | 0 | 0
  Week 3: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. |  |
  Week 23: Day 2: number analyzed (Participants) | 2 | 1 | 0
  Week 23: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. | 5.67 (NA) — SD was not estimable for a single participant. |
  Month 19: Day 2: number analyzed (Participants) | 0 | 3 | 2
  Month 19: Day 2 |  | 3.59 (0.763) | 6.61 (3.295)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 1
  Month 31: Day 2 |  | 4.80 (2.667) | 6.29 (NA) — SD was not estimable for a single participant.
  Month 43: number analyzed (Participants) | 0 | 4 | 2
  Month 43 |  | 4.33 (0.377) | 6.92 (1.154)
  Month 55: number analyzed (Participants) | 0 | 3 | 2
  Month 55 |  | 6.33 (1.548) | 8.25 (0.191)
  Month 67: number analyzed (Participants) | 0 | 2 | 2
  Month 67 |  | 6.10 (0.619) | 9.46 (2.319)
  Month 79: number analyzed (Participants) | 0 | 3 | 0
  Month 79 |  | 5.96 (2.207) |

14. Secondary Outcome: Volume of Distribution Associated With the Terminal Slope Following Extravascular Administration Divided by the Fraction of Dose Absorbed (Vz/F) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 6 | 5
liters
  Week 3: Day 2: number analyzed (Participants) | 3 | 0 | 0
  Week 3: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. |  |
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 0
  Week 23: Day 2 | 52.831 (NA) — SD was not estimable for a single participant. | 183.31 (NA) — SD was not estimable for a single participant. |
  Month 19: Day 2: number analyzed (Participants) | 0 | 3 | 2
  Month 19: Day 2 |  | 94.18 (21.961) | 152.82 (45.153)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 1
  Month 31: Day 2 |  | 116.91 (84.881) | 128.63 (NA) — SD was not estimable for a single participant.
  Month 43: number analyzed (Participants) | 0 | 4 | 2
  Month 43 |  | 68.06 (21.783) | 104.93 (44.848)
  Month 55: number analyzed (Participants) | 0 | 3 | 2
  Month 55 |  | 130.84 (15.624) | 127.77 (11.009)
  Month 67: number analyzed (Participants) | 0 | 2 | 2
  Month 67 |  | 115.31 (29.260) | 206.92 (11.864)
  Month 79: number analyzed (Participants) | 0 | 3 | 0
  Month 79 |  | 79.22 (8.364) |

15. Secondary Outcome: First Order Rate Constant (Lambda z) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: per hour (/h)
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 6 | 5
per hour (/h)
  Week 3: Day 2: number analyzed (Participants) | 3 | 0 | 0
  Week 3: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. |  |
  Week 23: Day 2: number analyzed (Participants) | 2 | 1 | 0
  Week 23: Day 2 | NA (NA) — Mean and SD were not estimable as values were below LLOQ. | 0.0309 (NA) — SD was not estimable for a single participant. |
  Month 19: Day 2: number analyzed (Participants) | 0 | 3 | 2
  Month 19: Day 2 |  | 0.0383 (0.00260) | 0.0419 (0.00917)
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 1
  Month 31: Day 2 |  | 0.0487 (0.01996) | 0.0489 (NA) — SD was not estimable for a single participant.
  Month 43: number analyzed (Participants) | 0 | 4 | 2
  Month 43 |  | 0.0677 (0.01829) | 0.0700 (0.01892)
  Month 55: number analyzed (Participants) | 0 | 3 | 2
  Month 55 |  | 0.0486 (0.01126) | 0.0649 (0.00708)
  Month 67: number analyzed (Participants) | 0 | 2 | 2
  Month 67 |  | 0.0539 (0.00831) | 0.0455 (0.00860)
  Month 79: number analyzed (Participants) | 0 | 3 | 0
  Month 79 |  | 0.0772 (0.03550) |

16. Secondary Outcome: Terminal Half-life (t1/2) of Idursulfase Administered as Intrathecal and in Conjunction With Elaprase
Description: Participants in 1 mg arm group were assessed for PK analysis in the HGT-HIT-045 study. T1/2 is calculated by dividing 0.693 by Lambda z. Here, 0.693 is the natural logarithm of 2 and Lambda z is the first order rate constant.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 3 | 6 | 5
hours
  Week 3: Day 2: number analyzed (Participants) | 3 | 0 | 0
  Week 3: Day 2 | NA [NA to NA] — Median and Full range were not estimable as values were below LLOQ. |  |
  Week 23: Day 2: number analyzed (Participants) | 1 | 1 | 0
  Week 23: Day 2 | NA [NA to NA] — T½ was not estimable due to non-availability of the Lambda z values. | 22.43 [NA to NA] — Full range was not estimable for a single participant. |
  Month 19: Day 2: number analyzed (Participants) | 0 | 3 | 2
  Month 19: Day 2 |  | 18.20 [16.9 to 19.4] | 16.94 [14.3 to 19.6]
  Month 31: Day 2: number analyzed (Participants) | 0 | 6 | 1
  Month 31: Day 2 |  | 15.57 [8.35 to 29.8] | 14.16 [NA to NA] — Full range was not estimable for a single participant.
  Month 43: number analyzed (Participants) | 0 | 4 | 2
  Month 43 |  | 10.28 [8.21 to 14.7] | 10.28 [8.31 to 12.2]
  Month 55: number analyzed (Participants) | 0 | 3 | 2
  Month 55 |  | 14.21 [11.6 to 18.6] | 10.75 [9.92 to 11.6]
  Month 67: number analyzed (Participants) | 0 | 2 | 2
  Month 67 |  | 13.01 [11.6 to 14.4] | 15.52 [13.4 to 17.6]
  Month 79: number analyzed (Participants) | 0 | 3 | 0
  Month 79 |  | 9.68 [6.02 to 15.4] |

17. Secondary Outcome: Total Body Clearance (CL) of Elaprase
Time Frame: 15 minutes prior to IV infusion, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 9, 11, and 24 hours during/after the IV infusion on Days 3-7 of Weeks 3 and 23
Population: Participants who received only Elaprase in HGT-HIT-045 and had evaluable samples were analyzed for this outcome measure. Number analyzed indicates the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: liters per hour (L/h)
Groups:
- Elaprase IV Infusion 0.5 mg/kg: Participants received 0.5 mg/kg SoC therapy of Elaprase IV infusions for up to a maximum of 157.2 months.
Arm/Group | Elaprase IV Infusion 0.5 mg/kg
Number analyzed (Participants) | 2
liters per hour (L/h)
  Week 3: Day 3-7 | 1.94 (1.677)
  Week 23: Day 3-7: number analyzed (Participants) | 1
  Week 23: Day 3-7 | 3.47 (NA) — SD was not estimable for a single participant.

18. Secondary Outcome: Observed Steady-state Volume of Distribution (Vss) of Elaprase
Time Frame: 15 minutes prior to IV infusion and at multiple timepoint (0.5, 1, 1.5, 2, 2.5, and 3 hours during the infusion; and at 3.5, 4, 5, 6, 7, 9, 11, and 24 hours) following IV infusion on Days 3-7 of Weeks 3 and 23
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Elaprase IV Infusion 0.5 mg/kg
Number analyzed (Participants) | 2
liters
  Week 3: Day 3-7 | 9.40 (3.464)
  Week 23: Day 3-7: number analyzed (Participants) | 1
  Week 23: Day 3-7 | 13.19 (NA) — SD was not estimable for a single participant.

19. Secondary Outcome: Volume of Distribution (Vz) of Elaprase
Description: Volume of distribution associated with the terminal slope (Vz) of Elaprase was assessed.
Time Frame: 15 minutes prior to IV infusion and at multiple timepoints (0.5, 1, 1.5, 2, 2.5, and 3 hours during the infusion; and at 3.5, 4, 5, 6, 7, 9, 11, and 24 hours) following IV infusion on Days 3-7 of Weeks 3 and 23
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Elaprase IV Infusion 0.5 mg/kg
Number analyzed (Participants) | 2
liters
  Week 3: Day 3-7 | 19.91 (13.874)
  Week 23: Day 3-7: number analyzed (Participants) | 1
  Week 23: Day 3-7 | 34.20 (NA) — SD was not estimable for a single participant.

20. Secondary Outcome: Mean Residence Time Extrapolated to Infinity (MRT0-inf) of Elaprase
Time Frame: as for outcome 19
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Elaprase IV Infusion 0.5 mg/kg
Number analyzed (Participants) | 2
hours
  Week 3: Day 3-7 | 6.49 (3.817)
  Week 23: Day 3-7: number analyzed (Participants) | 1
  Week 23: Day 3-7 | 3.80 (NA) — SD was not estimable for a single participant.

21. Secondary Outcome: Change From Baseline in CSF Biomarkers
Description: Change from baseline in CSF biomarkers glycosaminoglycan (GAG [heparan sulfate (HS)/dermatan sulfate (DS)]) was assessed.
Time Frame: Baseline, Months 7, 55, and 139
Population: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and have had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study. Number analyzed is the number of participants with data available for analyses. A few participants from the 1 mg arm had transitioned to 10 mg arm before the analysis at Month 7 was performed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
ng/mL
  Baseline: number analyzed (Participants) | 4 | 6 | 5
  Baseline | 1922.34 (1164.679) | 1874.00 (979.459) | 1111.92 (485.898)
  Change from Baseline at Month 7: number analyzed (Participants) | 2 | 7 | 5
  Change from Baseline at Month 7 | -807.50 (569.461) | -1526.24 (638.893) | -987.65 (437.885)
  Change from Baseline at Month 55: number analyzed (Participants) | 0 | 9 | 3
  Change from Baseline at Month 55 |  | -1575.63 (906.621) | -974.07 (558.075)
  Change from Baseline at Month 139: number analyzed (Participants) | 0 | 4 | 1
  Change from Baseline at Month 139 |  | -1169.25 (530.781) | -1135.51 (NA) — SD was not estimable for a single participant.

22. Secondary Outcome: Change From Baseline in Urinary Glycosaminoglycan (GAG)
Description: mg GAG/mmol creatinine stands for milligrams of GAG per millimole of creatinine.
Time Frame: Baseline, Months 7, 55, and 163
Population: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and have had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: mg GAG/mmol creatinine
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
Number analyzed (Participants) | 4 | 10 | 5
mg GAG/mmol creatinine
  Baseline: number analyzed (Participants) | 4 | 6 | 4
  Baseline | 34.07 (20.132) | 23.35 (13.799) | 13.67 (7.200)
  Change from Baseline at Month 7: number analyzed (Participants) | 4 | 6 | 3
  Change from Baseline at Month 7 | 5.22 (6.084) | -4.20 (4.278) | 3.35 (1.324)
  Change from Baseline at Month 55: number analyzed (Participants) | 0 | 7 | 3
  Change from Baseline at Month 55 |  | -6.83 (5.837) | 6.33 (7.387)
  Change from Baseline at Month 163: number analyzed (Participants) | 0 | 2 | 0
  Change from Baseline at Month 163 |  | -13.88 (5.163) |

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to 165 months)
Description: Safety Population included all eligible participants from HGT-HIT-045 who had agreed to participate in the extension study and have had either surgical implantation of an IDDD or intrathecal administration of study drug in the extension study. For Idursulfase-IT 1 mg+10 mg arm the AEs includes only the AEs that occurred while the participants were assigned to 10 mg.
Arm/Group | Idursulfase-IT 1 mg | Idursulfase-IT 10 mg | Idursulfase-IT 30 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/4 | 9/10 | 4/5
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idursulfase-IT 1 mg (N=4) | Idursulfase-IT 10 mg (N=10) | Idursulfase-IT 30 mg (N=5)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Atonic seizures (Nervous system disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CSF white blood cell count increased (Investigations) | 0 | 0 | 1
Central nervous system infection (Infections and infestations) | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 3 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Device breakage (General disorders) | 1 | 4 | 1
Device connection issue (General disorders) | 0 | 1 | 0
Device difficult to use (General disorders) | 1 | 0 | 0
Device dislocation (General disorders) | 1 | 4 | 0
Device failure (General disorders) | 0 | 5 | 2
Device malfunction (General disorders) | 1 | 4 | 2
Device occlusion (General disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Granuloma (General disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0 | 2
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Overgrowth bacterial (Infections and infestations) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 0
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 1 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular complication associated with device (General disorders) | 0 | 3 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idursulfase-IT 1 mg (N=4) | Idursulfase-IT 10 mg (N=10) | Idursulfase-IT 30 mg (N=5)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 2 | 0
Aggression (Psychiatric disorders) | 2 | 3 | 3
Agitation (Psychiatric disorders) | 1 | 8 | 3
Agitation postoperative (Injury, poisoning and procedural complications) | 0 | 5 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 2
Angiokeratoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anisocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0
Anticipatory anxiety (Psychiatric disorders) | 0 | 0 | 1
Antisocial behaviour (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 2 | 1
Application site erythema (General disorders) | 0 | 1 | 0
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Asthenia (General disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0
Bacterial test (Investigations) | 0 | 3 | 0
Bacterial test positive (Investigations) | 0 | 1 | 0
Bacterial tracheitis (Infections and infestations) | 0 | 1 | 0
Band neutrophil count increased (Investigations) | 0 | 2 | 0
Base excess decreased (Investigations) | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 2 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Blood calcium decreased (Investigations) | 0 | 2 | 1
Blood chloride increased (Investigations) | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Blood lactic acid increased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 0
Blood pressure decreased (Investigations) | 2 | 7 | 2
Blood pressure diastolic decreased (Investigations) | 2 | 8 | 2
Blood pressure diastolic increased (Investigations) | 1 | 8 | 2
Blood pressure fluctuation (Vascular disorders) | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 6 | 1
Blood pressure systolic decreased (Investigations) | 2 | 7 | 2
Blood pressure systolic increased (Investigations) | 2 | 8 | 2
Blood sodium increased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 3 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1
Bloody discharge (Vascular disorders) | 0 | 1 | 0
Body temperature decreased (Investigations) | 1 | 6 | 2
Body temperature increased (Investigations) | 1 | 2 | 2
Bone density decreased (Investigations) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 0
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bruxism (Psychiatric disorders) | 0 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
CSF cell count increased (Investigations) | 1 | 7 | 1
CSF culture positive (Investigations) | 0 | 0 | 1
CSF glucose decreased (Investigations) | 0 | 4 | 2
CSF lymphocyte count increased (Investigations) | 0 | 1 | 0
CSF neutrophil count positive (Investigations) | 0 | 0 | 1
CSF protein decreased (Investigations) | 0 | 1 | 0
CSF protein increased (Investigations) | 1 | 7 | 3
CSF white blood cell count increased (Investigations) | 1 | 0 | 0
Candida nappy rash (Infections and infestations) | 0 | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 4 | 4
Carpal tunnel syndrome (Nervous system disorders) | 0 | 5 | 3
Catheter site bruise (General disorders) | 1 | 0 | 1
Catheter site erythema (General disorders) | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 2 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 6 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 1
Chills (General disorders) | 0 | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Clonus (Nervous system disorders) | 1 | 2 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Congenital bowing of long bones (Congenital, familial and genetic disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 4 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 7 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 8 | 3
Convulsion (Nervous system disorders) | 0 | 6 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 3 | 0
Coronavirus test positive (Investigations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 8 | 3
Crepitations (General disorders) | 0 | 0 | 1
Croup infectious (Infections and infestations) | 0 | 1 | 1
Crystal urine present (Investigations) | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1 | 1
Cyst (General disorders) | 0 | 1 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Decreased activity (Psychiatric disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 6 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Device breakage (General disorders) | 0 | 3 | 0
Device connection issue (General disorders) | 0 | 1 | 0
Device dislocation (General disorders) | 0 | 2 | 0
Device malfunction (General disorders) | 1 | 4 | 1
Device occlusion (General disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 3
Discomfort (General disorders) | 0 | 2 | 0
Drooling (Nervous system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Dyskinesia (Nervous system disorders) | 1 | 1 | 0
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 1
Dysphemia (Psychiatric disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 2 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 7 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0
Eating disorder (Psychiatric disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema eyelids (Eye disorders) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 3 | 1
Electroencephalogram abnormal (Investigations) | 0 | 1 | 0
Energy increased (General disorders) | 0 | 1 | 0
Enterobiasis (Infections and infestations) | 1 | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 3
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 7 | 4
Exposure via ingestion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Extravasation (General disorders) | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 2 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 1
Eyelid margin crusting (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 6 | 4
Fatigue (General disorders) | 0 | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 3 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 2 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0
Gait disturbance (General disorders) | 2 | 6 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 4 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1
Generalised oedema (General disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 4 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 4 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 4 | 2
Heart rate decreased (Investigations) | 2 | 8 | 2
Heart rate increased (Investigations) | 0 | 4 | 1
Heart rate irregular (Investigations) | 0 | 0 | 1
Heart sounds abnormal (Investigations) | 1 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 1
Human bite (Injury, poisoning and procedural complications) | 0 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 3 | 2
Hypertonia (Nervous system disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochromasia (Blood and lymphatic system disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 4 | 3
Hypothermia (General disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 1
Implant site effusion (General disorders) | 1 | 4 | 0
Implant site erythema (General disorders) | 1 | 1 | 2
Implant site infection (Infections and infestations) | 0 | 0 | 1
Implant site pain (General disorders) | 0 | 1 | 0
Implant site rash (General disorders) | 0 | 0 | 1
Implant site reaction (General disorders) | 0 | 1 | 0
Implant site scar (General disorders) | 1 | 0 | 0
Implant site swelling (General disorders) | 0 | 4 | 1
Impulsive behaviour (Psychiatric disorders) | 0 | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 3 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion site bruising (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 3 | 3
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3 | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 3
Iron binding capacity total decreased (Investigations) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 4 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 3 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 1 | 0
Left atrial hypertrophy (Cardiac disorders) | 0 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 3 | 0
Leukocyte vacuolisation (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lice infestation (Infections and infestations) | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 1
Local swelling (General disorders) | 0 | 4 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Lymphocyte morphology abnormal (Investigations) | 0 | 1 | 0
Macrogenia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 3 | 2
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mastoid disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Mastoid effusion (Ear and labyrinth disorders) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 1 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 1 | 0
Mean cell volume abnormal (Investigations) | 0 | 1 | 0
Mean cell volume decreased (Investigations) | 0 | 4 | 0
Medical device complication (General disorders) | 1 | 1 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Microcytosis (Blood and lymphatic system disorders) | 0 | 3 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 3 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0
Monocyte morphology abnormal (Investigations) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0
Movement disorder (Nervous system disorders) | 0 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal odour (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasogastric output abnormal (Investigations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 8 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Negativism (Psychiatric disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 0
Nitrite urine present (Investigations) | 0 | 2 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 0 | 1 | 0
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 2 | 1
Otitis media (Infections and infestations) | 1 | 5 | 2
Otitis media acute (Infections and infestations) | 0 | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 5 | 2
Oxygen saturation decreased (Investigations) | 0 | 7 | 2
PCO2 decreased (Investigations) | 0 | 0 | 1
Pain (General disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3
Pallor (Vascular disorders) | 0 | 2 | 1
Papilloedema (Eye disorders) | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Parkinsonian gait (Nervous system disorders) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2
Penile erythema (Reproductive system and breast disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pica (Metabolism and nutrition disorders) | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 4 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 2
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 2
Procedural complication (Injury, poisoning and procedural complications) | 1 | 2 | 2
Procedural headache (Injury, poisoning and procedural complications) | 0 | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 4 | 2
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 8 | 5
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 3 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 3 | 2
Protein total increased (Investigations) | 0 | 1 | 0
Protein urine (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Protrusion tongue (Gastrointestinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pseudomonas test positive (Investigations) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 2 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Punctate basophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 0 | 1
Pupils unequal (Eye disorders) | 0 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 9 | 5
Radiculopathy (Nervous system disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 7 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 4 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Red blood cell burr cells present (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 2 | 0
Red blood cell count increased (Investigations) | 0 | 1 | 0
Red blood cells CSF positive (Investigations) | 1 | 2 | 1
Red blood cells urine (Investigations) | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 2 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Regressive behaviour (Psychiatric disorders) | 0 | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory rate decreased (Investigations) | 0 | 2 | 0
Respiratory rate increased (Investigations) | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 5 | 0
Retching (Gastrointestinal disorders) | 0 | 2 | 0
Retinal deposits (Eye disorders) | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 3 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 3
Rhinovirus infection (Infections and infestations) | 0 | 3 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Right ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scarlet fever (Infections and infestations) | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 3 | 3
Seasonal allergy (Immune system disorders) | 1 | 3 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 5 | 1
Skin candida (Infections and infestations) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Skull malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 3 | 1
Sleep study abnormal (Investigations) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Social avoidant behaviour (Psychiatric disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Splinter (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Staring (Psychiatric disorders) | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thirst (General disorders) | 0 | 1 | 1
Thyroid function test abnormal (Investigations) | 0 | 0 | 1
Thyroxine decreased (Investigations) | 0 | 1 | 0
Thyroxine increased (Investigations) | 0 | 3 | 0
Tinea pedis (Infections and infestations) | 0 | 2 | 2
Toe walking (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1
Tooth abscess (Infections and infestations) | 0 | 2 | 1
Tooth crowding (Gastrointestinal disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 1 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Transferrin decreased (Investigations) | 0 | 1 | 0
Transferrin saturation increased (Investigations) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic lumbar puncture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 2 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 1 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 8 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 1 | 0
Urobilinogen urine increased (Investigations) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Vascular complication associated with device (General disorders) | 1 | 7 | 5
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 10 | 4
Weight decreased (Investigations) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Xanthochromia (Investigations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT01506141/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT01506141/SAP_001.pdf